CLINICAL TRIAL: NCT03572218
Title: A Randomized Controlled Trial of a Psychological Intervention to Reduce Weight Bias Internalization in the Context of Behavioral Weight Loss
Brief Title: Psychological Intervention to Reduce Weight Bias Internalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Rebecca L. Pearl, Ph.D., Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 829070
Record Dates: First submitted 2018-06-04; First posted 2018-06-28 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Stigmatization; Obesity; Weight Loss
MeSH Terms: conditions — Stereotyping; Obesity; Weight Loss | interventions — Bias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWL + BIAS (Experimental): The behavioral weight loss (BWL) + weight bias internalization and stigma (BIAS) group will include standard BWL treatment (described in more detail in Intervention section) combined with a weight stigma-reduction intervention. During the initial 12 weeks, the weekly 60-minute BWL sessions will be followed by 30 minutes devoted to stigma-related content. In the every-other-week and monthly weight loss maintenance sessions from weeks 13-26, strategies for coping with weight stigma and challenging internalized beliefs will be reviewed, and participants will be encouraged to use these strategies specifically in the context of weight management.
  Interventions: Behavioral: BWL; Behavioral: BIAS
- Standard BWL (Active Comparator): The Standard BWL group will receive weekly BWL sessions (described in more detail in Intervention section) for 12 weeks, followed by every-other-week and monthly weight loss maintenance sessions from weeks 13-26. BWL content will last for 60 minutes, with an additional 30 minutes in this group devoted to discussing recipes and food preparation.
  Interventions: Behavioral: BWL

INTERVENTIONS:
Behavioral: BWL — The BWL sessions will be based on the Diabetes Prevention Program (DPP) manual. A diet of 1200-1499 calories per day will be prescribed for participants < 250 lb, and 1500-1800 for those ≥ 250 lb. Participants will be instructed to eat a balanced deficit diet. Session topics during the first 12 weeks will include self-monitoring, stimulus control, slowing eating, social support, cognitive restructuring, portion sizes, and goal-setting. Those during weeks 13-26 will focus on continued self-monitoring and skills required for weight loss maintenance and relapse prevention. Physical activity will be prescribed at a level consistent with data showing that >250 min/wk is associated with improved long-term weight loss. BWL sessions will last 60 minutes.
Behavioral: BIAS — Following 60 minutes of BWL treatment, the BIAS intervention will devote 30 minutes to stigma-related content. Session topics will include: psychoeducation about weight and weight stigma; challenging myths and cognitive distortions related to weight; strategies for coping with instances of stigma; and increasing empowerment and body esteem. The effects of weight stigma on health behaviors will be discussed, and sessions will focus specifically on helping participants overcome stigma-related barriers to weight management. In the every-other-week and monthly weight loss maintenance sessions from weeks 13-26, strategies for coping with weight stigma and challenging internalized beliefs will be reviewed, and participants will be encouraged to use these strategies in the context of weight management.
  Arms: BWL + BIAS

SUMMARY:
This is a randomized controlled trial to test the effects on WBI of a novel psychological intervention combined with standard behavioral weight loss (BWL) treatment, as compared to BWL alone. Participants will be a total of 72 men and women seeking weight loss, ages 18-65 years, with a body mass index (BMI) of 30 kg/m2 or above, a history of experiencing weight bias, and elevated levels of WBI. Participants will attend a screening visit in which they will complete a behavioral evaluation with a psychologist and a medical history that will be reviewed by a nurse practitioner or physician. Questionnaires assessing experiences and internalization of weight bias, with confirmation by interviewer assessment during the behavioral evaluation, will be used to determine whether participants meet criteria for having high levels of WBI. Eligible consenting participants will be randomly assigned to the standard BWL intervention (n = 36) or the BWL + BIAS program (n = 36). All participants will attend weekly, 90-minute group meetings for 12 weeks (12 visits). In the BWL + stigma intervention, 60 minutes will be devoted to BWL and 30 minutes to weight stigma. In the standard BWL treatment group, the additional 30 minutes will be devoted to sharing recipes and food preparation tips. Following 12 weeks of weight loss treatment, participants will attend group meetings focused on weight loss maintenance, every-other-week from weeks 13-16 (2 visits), and monthly from weeks 17-26 (2 visits). Maintenance sessions in the BWL + stigma group will continue to incorporate discussion of WBI. Assessments - which include questionnaires and measurements of body weight - will occur at baseline and weeks 12 and 26. Weight will be measured at every group meeting for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be men and women ages 18-65 years.
* Participants must have obesity (defined as a BMI ≥ 30 kg/m2); report a history of experiencing weight bias as assessed by self-report questionnaire and in-person interview; and have elevated levels of WBI as indicated by an average score of 4 (midpoint) or above on the Weight Bias Internalization Scale (WBIS) and by in-person interview.
* Participants must be seeking weight loss.
* If currently taking medications, dosages must be stable for at least 3 months.
* Participants will be eligible to participate if they exhibit mild to moderate severity of depression, anxiety, or binge eating disorder, as determined by the behavioral evaluation and the screening measures (Beck Depression Inventory-II and Questionnaire for Eating and Weight Patterns; see below for details). Elevated WBIS scores are often associated with these variables.
* Participants taking anti-depressant medication will be eligible if their dose has been stable for a minimum of 3 months.

Eligible female patients will be:

* non-pregnant, evidenced by a negative urine dipstick pregnancy test
* non-lactating
* surgically sterile or postmenopausal, or they will agree to continue to use a method of birth control during the study

Participants must:

* have a PCP who is responsible for providing routine care
* have reliable telephone service with which to participate in conference calls
* understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent

Exclusion Criteria:

Applicants will be excluded if they have:

* a diagnosis of type I or II diabetes;
* uncontrolled hypertension (blood pressure ≥ 160/100 mm Hg);
* experienced a cardiovascular event (e.g., stroke, myocardial infarction) in the last 12 months;
* lost ≥ 5% of their initial weight in the last 6 months;
* or have participated in individual or group psychotherapy in the last 3 months (due to the potentially confounding effects of receiving a simultaneous cognitive-behavioral intervention). Applicants who have recently participated in or are currently receiving counseling for concerns unrelated to mood, self-esteem, or weight (e.g. career, marriage, or grief counseling; caregiver support) may be eligible per Principal Investigator's discretion.
* Applicants with severe symptoms of mood (for example, BDI-II score ≥ 29), anxiety, or binge eating disorder, and any severity of thought or substance use disorders will not be accepted into the study, as these symptoms may interfere with individuals' ability to adhere to a weight loss program. Clinician judgment will be used to determine severity of mood disorder symptoms independent from obesity-related concerns and complications (e.g., fatigue), and decisions about applicants' eligibility based on psychiatric symptoms will fall within the Principal Investigator's discretion.
* Individuals with bulimia nervosa will not be eligible to participate, because weight loss may be contraindicated.
* Applicants with current, active suicidal ideation, and/or a suicide attempt within the past year will be excluded from the study and referred to psychiatric treatment facilities in the greater Philadelphia area.
* Applicants will not be eligible if they have a history of bariatric surgery.
* Women who are nursing, pregnant, or planning to become pregnant in the next 12 months are not eligible to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Pearl, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- The University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Pearl RL, Wadden TA, Bach C, Tronieri JS, Berkowitz RI. Six-Month Follow-up from a Randomized Controlled Trial of the Weight BIAS Program. Obesity (Silver Spring). 2020 Oct;28(10):1878-1888. doi: 10.1002/oby.22931. Epub 2020 Aug 28. PMID 32860344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began April 2018 and ended October 2018. Participants were recruited by flyers, local media, and physician referrals for a study about weight loss and social experiences related to weight. Participants were screened by telephone and by a subsequent in-person behavioral evaluation and brief medical evaluation.
Groups:
- BWL + BIAS: In the behavioral weight loss (BWL) + weight bias internalization and stigma (BIAS) group, participants received 60-minute BWL sessions followed by 30 minutes of a weight stigma-reduction intervention. Participants received weekly group treatment sessions for 12 weeks, followed by every-other-week and monthly sessions from weeks 13-26.
- Standard BWL: In the BWL group, participants received 60-minute BWL sessions followed by 30 minutes devoted to discussing recipes and food preparation. Participants received weekly group treatment sessions for 12 weeks, followed by every-other-week and monthly sessions from weeks 13-26.
Period: Overall Study
Arm/Group | BWL + BIAS | Standard BWL
Started | 36 | 36
Week 12 | 30 | 31
Week 26 | 30 | 31
Completed | 30 | 31
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 3 | 2
Not completed — No longer available for study visits | 2 | 1
Not completed — No longer interested | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BWL + BIAS | Standard BWL | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (11.4) | 46.6 (11.8) | 47.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 22 | 48
  White | 7 | 14 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] — Average of duplicate measures of weight (with a digital scale; Detecto, model 6800A) obtained at baseline.
  kilograms | 112.4 (24.0) | 107.2 (21.2) | 109.8 (22.6)
Height [Mean (Standard Deviation); unit: centimeters] — Average of duplicate measures of height (with a wall-mounted stadiometer; Veeder-Root, Elizabethtown, NC) obtained at screening.
  centimeters | 167.0 (8.7) | 166.6 (8.5) | 166.8 (8.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated at baseline by dividing participants' baseline weight (kilograms, kg) by their screening height (meters, m) squared (kg/m^2).
  kg/m^2 | 40.1 (6.5) | 38.4 (5.6) | 39.3 (6.1)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] — Average of duplicate measures of waist circumference measured (to the nearest 0.1 centimeter) with flexible tension-controlled measuring tape midway between the iliac crest and lowest rib.
  centimeters | 119.1 (15.3) | 114.9 (12.6) | 117.0 (14.1)
Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Average of duplicate measures of blood pressure (systolic blood pressure and diastolic blood pressure; mmHg) obtained at screening using an automated Dinamap monitor (Johnson & Johnson, XL model 9300) at 1-minute intervals after ≥ 5 minute rest, controlling for blood pressure medication
  mmHg
    Systolic Blood Pressure | 127.4 (10.2) | 128.0 (10.7) | 127.7 (10.3)
    Diastolic Blood Pressure | 73.0 (9.2) | 74.3 (7.9) | 73.7 (8.5)
Weight Bias Internalization [Mean (Standard Deviation); unit: scores on a scale] — The Weight Bias Internalization Scale assesses weight bias internalization. Average of 11 items, rated 1-7 (higher scores indicate higher weight bias internalization)
  scores on a scale | 5.0 (0.7) | 5.2 (0.7) | 5.1 (0.7)
Weight Self-Stigma Questionnaire (WSSQ) [Mean (Standard Deviation); unit: scores on a scale] — Sum of 12 items (WSSQ-Total; rated 1-5). The WSSQ consists of two subscales: Self-Devaluation (WSSQ-SD; 6 items) and Fear of Enacted Stigma (WSSQ-FNE; 6 items); higher scores indicate greater weight self-stigma. Population: All participants who completed the questionnaires assessing secondary outcomes at baseline.
  scores on a scale
    WSSQ-Total: number analyzed (Participants) | 36 | 35 | 71
    WSSQ-Total | 37.9 (6.6) | 39.3 (6.9) | 38.6 (6.7)
    WSSQ-SD: number analyzed (Participants) | 36 | 35 | 71
    WSSQ-SD | 19.1 (4.2) | 19.2 (3.9) | 19.2 (4.1)
    WSSQ-FNE: number analyzed (Participants) | 36 | 35 | 71
    WSSQ-FNE | 18.8 (4.6) | 20.1 (4.8) | 19.4 (4.7)
Weight Bias [Mean (Standard Deviation); unit: scores on a scale] — The Fat Phobia Scale assesses weight bias. Participants rated 14 pairs of adjectives used to describe people with obesity using a differential rating scale (1-5) to indicate whether or not they agreed with negative weight stereotypes. Scores are averaged 1-5, with higher scores indicating greater weight bias. Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 3.7 (0.7) | 3.7 (0.6) | 3.7 (0.6)
Depression [Mean (Standard Deviation); unit: scores on a scale] — The Patient Health Questionnaire-9 assesses symptoms of depression. Sum of 9 items, rated 0-3. Scores range from 0-27 (higher scores indicate more symptoms of depression). Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 7.5 (5.1) | 8.4 (4.5) | 8.0 (4.8)
Anxiety [Mean (Standard Deviation); unit: scores on a scale] — The Generalized Anxiety Disorder-7 Questionnaire assesses anxiety. Sum of 7 items, rated 0-3. Scores range from 0-21 (higher scores indicate greater anxiety). Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 5.6 (4.5) | 5.2 (4.2) | 5.4 (4.3)
Perceived Stress [Mean (Standard Deviation); unit: scores on a scale] — The Perceived Stress Scale assesses self-reported daily stress. Sum of 10 items, rated 0-4. Total scores range from 0-40 (higher scores indicate greater perceived stress). Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 17.6 (6.2) | 16.9 (6.5) | 17.3 (6.4)
Body Esteem [Mean (Standard Deviation); unit: scores on a scale] — The Body Appreciation Scale assesses body esteem. Average of 10 items (rated 1-5; higher scores indicate greater body appreciation) Population: All participants who completed the questionnaires assessing secondary outcome at baseline
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 2.8 (0.6) | 2.5 (0.7) | 2.6 (0.7)
Weight-Related Quality of Life [Mean (Standard Deviation); unit: scores on a scale] — The Impact of Weight on Quality of Life Questionnaire- Lite assess weight-related quality of life. Sum of 31 items (containing 5 subscales; rated 1-5) used to assess weight-specific aspects of psychological and physical functioning. Scores transformed to a 0-100 scale, with higher scores indicating better quality of life. Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 56.3 (16.7) | 54.2 (16.5) | 55.3 (16.5)
Eating Self-Efficacy [Mean (Standard Deviation); unit: scores on a scale] — The Weight and Lifestyle Efficacy - Short Form assesses confidence in one's ability to overcome challenges that lead to overeating. Sum of 8 items (rated 0-10). Total scores range from 0-80 (higher scores indicate greater self-efficacy). Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 39.4 (17.4) | 40.7 (17.9) | 40.0 (17.5)
Exercise Self-Efficacy [Mean (Standard Deviation); unit: scores on a scale] — The Self-Efficacy for Exercise Scale assesses confidence to overcome barriers to physical activity. Sum of 9 items (rated 0-10). Total scores range from 0-90 (higher scores indicate greater exercise self-efficacy). Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    number analyzed (Participants) | 36 | 35 | 71
    (all) | 48.3 (20.1) | 54.2 (19.9) | 51.2 (20.0)
Eating Behaviors [Mean (Standard Deviation); unit: scores on a scale] — The Eating Inventory Questionnaires assesses eating behaviors and consists of subscales: Dietary Restraint (21 items), Disinhibition (16 items), and Hunger (14 items). Items include both true/false statements and rating scales, with all scores converted to 0 or 1 ratings and summed. Higher scores indicate greater restraint/disinhibition/hunger. Population: All participants who completed the questionnaires assessing secondary outcomes at baseline.
  scores on a scale
    Dietary Restraint: number analyzed (Participants) | 36 | 35 | 71
    Dietary Restraint | 8.5 (3.7) | 8.9 (3.8) | 8.7 (3.7)
    Disinhibition: number analyzed (Participants) | 36 | 35 | 71
    Disinhibition | 9.2 (3.5) | 10.2 (3.1) | 9.7 (3.3)
    Hunger: number analyzed (Participants) | 36 | 35 | 71
    Hunger | 7.8 (3.6) | 6.4 (3.6) | 7.1 (3.7)
Self-Reported Self-Monitoring Behaviors [Mean (Standard Deviation); unit: scores on a scale] — Rated frequency of self-monitoring for: Self-Reported Weighing (rated 0-4, less than once per month through several times per day), Track Food/Drink (rated 0-4, from never to everyday), Track Calories (rated 0-4, from never to everyday), and Track Activity (rated 0-4, from never to everyday) Population: All participants who completed the questionnaires assessing secondary outcome at baseline.
  scores on a scale
    Self-Reported Weighing: number analyzed (Participants) | 36 | 35 | 71
    Self-Reported Weighing | 0.9 (1.2) | 0.9 (1.1) | 0.9 (1.2)
    Track Food/Drink: number analyzed (Participants) | 36 | 35 | 71
    Track Food/Drink | 0.4 (0.7) | 0.5 (0.8) | 0.5 (0.8)
    Track Calories: number analyzed (Participants) | 36 | 35 | 71
    Track Calories | 0.4 (1.0) | 0.6 (1.1) | 0.5 (1.0)
    Track Activity: number analyzed (Participants) | 36 | 35 | 71
    Track Activity | 1.0 (1.5) | 1.3 (1.5) | 1.2 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Weight Bias Internalization
Description: Estimated mean change score on the Weight Bias Internalization Scale (scale scoring 1-7; higher scores indicate greater weight bias internalization)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -1.3 (0.2) | -1.0 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.2

2. Secondary Outcome: Weight Bias Internalization
Description: as for outcome 1
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -1.5 (0.2) | -1.3 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.3

3. Secondary Outcome: Weight Self-Stigma Questionnaire (WSSQ)
Description: Estimated mean change score for Total score (WSSQ-Total, summed 12-60) and two subscales of Self-Devaluation (WSSQ-SD) and Fear of Enacted Stigma (WSSQ-FNE) (summed 6-30); higher scores indicate greater weight self-stigma
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  WSSQ-Total | -6.0 (1.4) | -1.6 (1.3)
  WSSQ-SD | -3.6 (0.8) | -1.0 (0.8)
  WSSQ-FNE | -2.3 (0.8) | -0.7 (0.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; WSSQ-Total; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -4.4, Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; WSSQ-SD; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -2.8, Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; WSSQ-FNE; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = -1.6, Standard Error of Mean 1.2

4. Secondary Outcome: Weight Self-Stigma Questionnaire (WSSQ)
Description: as for outcome 3
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  WSSQ-Total | -7.1 (1.5) | -3.6 (1.5)
  WSSQ-SD | -4.1 (0.8) | -1.5 (0.8)
  WSSQ-FNE | -2.9 (0.9) | -2.1 (0.9)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; WSSQ-Total; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -3.5, Standard Error of Mean 2.1
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; WSSQ-SD; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = -2.6, Standard Error of Mean 1.1
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; WSSQ-FNE; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = -0.8, Standard Error of Mean 1.3

5. Secondary Outcome: Weight Bias
Description: Estimated mean change score on the Fat Phobia Scale (scale scoring 1-5; higher scores indicate greater weight bias)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -0.5 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.2

6. Secondary Outcome: Weight Bias
Description: Estimated mean change score on the Fat Phobia Scale (scale scoring 1-5; higher scores indicate greater weight bias)
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -0.5 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.2

7. Secondary Outcome: Weight-Related Quality of Life
Description: Estimated mean change score on the Impact of Weight on Quality of Life Questionnaire-Lite for Total score and five subscales of Physical Function, Self Esteem, Sexual Life, Work, and Public Distress (transformed scores 0-100; higher scores indicate better quality of life)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Total | 8.3 (2.1) | 8.9 (2.0)
  Physical Function | 9.8 (2.9) | 8.8 (2.8)
  Self Esteem | 12.9 (3.0) | 9.2 (3.0)
  Sexual Life | 5.5 (3.6) | 9.5 (3.5)
  Work | 4.8 (3.1) | 6.9 (3.0)
  Public Distress | 5.7 (2.6) | 7.7 (2.6)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Impact of Weight on Quality of Life Questionnaire-Lite for Total score; Test type: Superiority; p = 0.84, Mixed Models Analysis; Mean Difference (Net) = -0.6, Standard Error of Mean 2.9
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Physical Function Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = 0.9, Standard Error of Mean 4.0
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Self Esteem Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.39, Mixed Models Analysis; Mean Difference (Net) = 3.7, Standard Error of Mean 4.3
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Sexual Life Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = -4.0, Standard Error of Mean 5.0
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Work Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Net) = -2.0, Standard Error of Mean 4.3
Statistical Analysis 6: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Public Distress Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Net) = -2.0, Standard Error of Mean 3.6

8. Secondary Outcome: Weight-Related Quality of Life
Description: as for outcome 7
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Total | 12.5 (2.1) | 14.1 (2.1)
  Physical Function | 13.7 (2.9) | 14.2 (2.8)
  Self Esteem | 19.1 (3.4) | 18.5 (3.3)
  Sexual Life | 7.0 (3.6) | 14.0 (3.5)
  Work | 8.6 (3.1) | 6.8 (3.0)
  Public Distress | 9.9 (2.6) | 11.2 (2.6)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Impact of Weight on Quality of Life Questionnaire-Lite for Total score; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Net) = -1.7, Standard Error of Mean 3.0
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Net) = -0.5, Standard Error of Mean 4.0
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Self Esteem Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.90, Mixed Models Analysis; Mean Difference (Net) = 0.6, Standard Error of Mean 4.7
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Sexual Life Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = -7.1, Standard Error of Mean 5.0
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Estimated mean change score on the Work Subscale of the Impact of Weight on Quality of Life Questionnaire-Lite; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Net) = 1.8, Standard Error of Mean 4.3
Statistical Analysis 6: Comparison: BWL + BIAS vs Standard BWL; [analysis description as in outcome 7, analysis 6]; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Net) = -1.3, Standard Error of Mean 3.6

9. Secondary Outcome: Perceived Stress
Description: Estimated mean change score on the Perceived Stress Scale (summed 0-40; higher scores indicate greater perceived stress)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -3.2 (1.2) | -0.1 (1.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Net) = -3.0, Standard Error of Mean 1.7

10. Secondary Outcome: Perceived Stress
Description: as for outcome 9
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -3.9 (1.2) | -1.0 (1.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.10, Mixed Models Analysis; Mean Difference (Net) = -2.9, Standard Error of Mean 1.7

11. Secondary Outcome: Depression
Description: Estimated mean change score on the Patient Health Questionnaire - 9 (summed 0-27; higher scores indicate more symptoms of depression)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -3.4 (0.8) | -2.5 (0.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Net) = -0.9, Standard Error of Mean 1.1

12. Secondary Outcome: Depression
Description: as for outcome 11
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -2.9 (0.8) | -2.9 (0.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.98, Mixed Models Analysis; Mean Difference (Net) = -0.03, Standard Error of Mean 1.1

13. Secondary Outcome: Exercise Self-Efficacy
Description: Estimated mean change score on the Self-Efficacy for Exercise Scale (summed 0-90; higher scores indicate greater self-efficacy)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 4.0 (4.6) | -5.7 (4.5)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = 9.7, Standard Error of Mean 6.5

14. Secondary Outcome: Exercise Self-Efficacy
Description: as for outcome 13
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 5.8 (4.6) | -6.3 (4.5)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.06, Mixed Models Analysis; Mean Difference (Net) = 12.1, Standard Error of Mean 6.5

15. Secondary Outcome: Eating Self-Efficacy
Description: Estimated mean change score on the Weight and Lifestyle Efficacy - Short Form (summed 0-80; higher scores indicate greater self-efficacy)
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 11.3 (3.1) | 10.2 (3.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Net) = 1.1, Standard Error of Mean 4.4

16. Secondary Outcome: Eating Self-Efficacy
Description: as for outcome 15
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 12.0 (3.1) | 8.9 (3.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = 3.1, Standard Error of Mean 4.4

17. Secondary Outcome: Percent Weight Change
Description: Estimated mean change in percent weight change. Weight measured in kilograms (kg).
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: percent weight change
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
percent weight change | -4.5 (1.0) | -5.9 (1.0)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Net) = 1.4, Standard Error of Mean 1.4

18. Secondary Outcome: Waist Circumference
Description: Estimated mean change in waist circumference (cm).
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: change in cm
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
change in cm | -4.3 (0.9) | -5.1 (0.9)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.54, Mixed Models Analysis; Mean Difference (Net) = 0.8, Standard Error of Mean 1.3

19. Secondary Outcome: Blood Pressure
Description: Estimated mean change in blood pressure (systolic blood pressure and diastolic blood pressure; mmHg), controlling for blood pressure medication.
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: change in mmHg
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
change in mmHg
  Systolic Blood Pressure | -2.6 (1.6) | -2.4 (1.6)
  Diastolic Blood Pressure | -1.5 (1.2) | -2.2 (1.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Systolic Blood Pressure; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 2.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Diastolic Blood Pressure; Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Net) = 0.8, Standard Error of Mean 1.6

20. Other Pre Specified Outcome: Coping Behaviors in Response to Weight Stigma
Description: Estimated mean change score on the Coping with Weight Stigma Questionnaire for Full scale and four subscales of Negative Affect, Maladaptive Eating, Healthy Lifestyle, and Exercise Avoidance (scale scoring 0-4 for Full scale and all subscales); higher scores indicate greater endorsement of coping strategies
Time Frame: Baseline to week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Full Scale | -0.7 (0.1) | -0.8 (0.1)
  Negative Affect | -1.1 (0.1) | -1.2 (0.1)
  Maladaptive Eating | -0.7 (0.1) | -0.7 (0.1)
  Healthy Lifestyle | 0.0 (0.2) | 0.1 (0.2)
  Exercise Avoidance | -0.8 (0.2) | -0.5 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Full Scale; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Negative Affect; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Maladaptive Eating; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Healthy Lifestyle; Test type: Superiority; p = 0.71, Mixed Models Analysis; Mean Difference (Net) = 0.2, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Exercise Avoidance; Test type: Superiority; p = 0.41, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.3

21. Other Pre Specified Outcome: Coping Behaviors in Response to Weight Stigma
Description: as for outcome 20
Time Frame: Baseline to week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Full Scale | -0.8 (0.1) | -0.9 (0.1)
  Negative Affect | -1.3 (0.2) | -1.2 (0.2)
  Maladaptive Eating | -0.8 (0.1) | -0.8 (0.1)
  Healthy Lifestyle | -0.2 (0.2) | 0.0 (0.2)
  Exercise Avoidance | -0.9 (0.2) | -0.9 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Full Scale; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Negative Affect; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Maladaptive Eating; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Healthy Lifestyle; Test type: Superiority; p = 0.47, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Exercise Avoidance; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 0.3

22. Other Pre Specified Outcome: Body Esteem
Description: Estimated mean change score on the Body Appreciation Scale (scale scoring 1-5; higher scores indicate greater body appreciation)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.6 (0.1) | 0.3 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.2

23. Other Pre Specified Outcome: Body Esteem
Description: as for outcome 22
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.8 (0.1) | 0.5 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.2

24. Other Pre Specified Outcome: Body Dissatisfaction
Description: Estimated mean change score on the Body Areas Satisfaction Subscale of the Multidimensional Body-Self Relations Questionnaire-Appearance Scales (scale scoring 1-5; higher scores indicating greater satisfaction)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.4 (0.1) | 0.4 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.1

25. Other Pre Specified Outcome: Body Dissatisfaction
Description: as for outcome 24
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.6 (0.1) | 0.5 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = 0.2, Standard Error of Mean 0.2

26. Other Pre Specified Outcome: Disordered Eating
Description: Estimated mean change score on the Eating Disorders Examination Questionnaire for Global score and four subscales of Eating Restraint, Eating Concern, Weight Concern, and Shape Concern (scale scoring 0-6 for Global score and all subscales; higher scores indicate greater pathology)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Global | -0.2 (0.1) | -0.2 (0.1)
  Eating Restraint | 1.7 (0.2) | 1.5 (0.2)
  Eating Concern | -0.4 (0.2) | -0.7 (0.2)
  Weight Concern | -0.7 (0.2) | -0.7 (0.2)
  Shape Concern | -1.1 (0.2) | -0.9 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Global; Test type: Superiority; p = 0.83, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Eating Restraint; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Eating Concern; Test type: Superiority; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Weight Concern; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Shape Concern; Test type: Superiority; p = 0.36, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.3

27. Other Pre Specified Outcome: Disordered Eating
Description: as for outcome 26
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Global | -0.5 (0.1) | -0.3 (0.1)
  Eating Restraint | 1.2 (0.2) | 1.0 (0.2)
  Eating Concern | -0.7 (0.2) | -0.6 (0.2)
  Weight Concern | -1.2 (0.2) | -0.8 (0.2)
  Shape Concern | -1.4 (0.2) | -1.0 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Global; Test type: Superiority; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Eating Restraint; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Eating Concern; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Weight Concern; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Net) = -0.4, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Shape Concern; Test type: Superiority; p = 0.18, Mixed Models Analysis; Mean Difference (Net) = -0.4, Standard Error of Mean 0.3

28. Other Pre Specified Outcome: Eating Behaviors
Description: Estimated mean change score on the Eating Inventory Questionnaire for three subscales of Dietary Restraint (summed 0-21), Disinhibition (summed 0-16), and Hunger (summed 0-14); higher values indicate greater restraint/disinhibition/hunger
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Dietary Restraint | 6.3 (0.7) | 5.9 (0.7)
  Disinhibition | -2.8 (0.6) | -1.9 (0.6)
  Hunger | -3.2 (0.5) | -1.4 (0.5)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Dietary Restraint; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Net) = 0.4, Standard Error of Mean 1.0
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Disinhibition; Test type: Superiority; p = 0.28, Mixed Models Analysis; Mean Difference (Net) = 0.9, Standard Error of Mean 0.8
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Hunger; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -1.8, Standard Error of Mean 0.8

29. Other Pre Specified Outcome: Eating Behaviors
Description: as for outcome 28
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Dietary Restraint | 6.4 (0.8) | 5.2 (0.8)
  Disinhibition | -3.0 (0.6) | -2.2 (0.6)
  Hunger | -3.9 (0.5) | -1.4 (0.5)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Dietary Restraint; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 1.2, Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Disinhibition; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mean Difference (Net) = -0.8, Standard Error of Mean 0.8
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Hunger; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -2.5, Standard Error of Mean 0.8

30. Other Pre Specified Outcome: Anxiety
Description: Estimated mean change score on the Generalized Anxiety Disorder-7 Questionnaire (summed 0-21; higher scores indicate greater anxiety)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -1.8 (0.8) | -0.7 (0.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Net) = -1.1, Standard Error of Mean 1.1

31. Other Pre Specified Outcome: Anxiety
Description: as for outcome 30
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -1.6 (0.8) | -0.8 (0.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = -0.8, Standard Error of Mean 1.2

32. Other Pre Specified Outcome: Dietary Monitoring
Description: Estimated mean change in number of days recording caloric intake
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: number of days
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
number of days | 52.9 (3.4) | 55.5 (3.4)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Net) = 2.6, Standard Error of Mean 4.8

33. Other Pre Specified Outcome: Dietary Monitoring
Description: Estimated mean change in number of days recording caloric intake
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: number of days
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
number of days | 85.6 (9.5) | 95.8 (9.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.44, Mixed Models Analysis; Mean Difference (Net) = -10.2, Standard Error of Mean 13.1

34. Other Pre Specified Outcome: Self-Reported Self-Monitoring Behaviors
Description: Estimated mean change in self-reported frequency of tracking of: weight, food/drink, calories, and physical activity; 0-4 rating for each of the four behaviors (higher scores indicate greater self-reported frequency of self-monitoring behavior)
Time Frame: Baseline to Week 12
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Self-Reported Weighing | 0.9 (0.2) | 1.1 (0.2)
  Track Food/Drink | 2.7 (0.3) | 2.0 (0.3)
  Track Calories | 2.0 (0.3) | 1.7 (0.3)
  Track Activity | 1.6 (0.3) | 0.8 (0.3)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Self-Reported Weighing; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Track Food/Drink; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Net) = 0.7, Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Track Calories; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Track Activity; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Net) = 0.8, Standard Error of Mean 0.4

35. Other Pre Specified Outcome: Self-Reported Self-Monitoring Behaviors
Description: as for outcome 34
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Self-Reported Weighing | 1.0 (0.2) | 0.6 (0.2)
  Track Food/Drink | 1.6 (0.3) | 1.6 (0.3)
  Track Calories | 1.7 (0.3) | 1.4 (0.3)
  Track Activity | 1.3 (0.3) | 0.9 (0.3)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Self-Reported Weighing; Test type: Superiority; p = 0.23, Mixed Models Analysis; Mean Difference (Net) = 0.4, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Track Food/Drink; Test type: Superiority; p = 0.90, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Track Calories; Test type: Superiority; p = 0.36, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Track Activity; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 0.5, Standard Error of Mean 0.4

36. Other Pre Specified Outcome: Weight Bias Internalization
Description: as for outcome 1
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale | -1.5 (0.2) | -1.2 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.3

37. Other Pre Specified Outcome: Weight Self-Stigma Questionnaire (WSSQ)
Description: as for outcome 3
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale
  WSSQ-Total | -5.6 (1.6) | -3.1 (1.6)
  WSSQ-SD | -2.9 (0.8) | -1.2 (0.8)
  WSSQ-FNE | -2.7 (1.0) | -2.0 (1.0)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; WSSQ-Total; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Net) = -2.5, Standard Error of Mean 2.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; WSSQ-SD; Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Net) = -1.8, Standard Error of Mean 1.2
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; WSSQ-FNE; Test type: Superiority; p = 0.65, Mixed Models Analysis; Mean Difference (Net) = 0.6, Standard Error of Mean 1.4

38. Other Pre Specified Outcome: Weight Bias
Description: Estimated mean change score on the Fat Phobia Scale (scale scoring 1-5; higher scores indicate greater weight bias)
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale | -0.4 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.21, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.2

39. Other Pre Specified Outcome: Depression
Description: as for outcome 11
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale | -2.9 (0.9) | -2.4 (0.9)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.7, Mixed Models Analysis; Mean Difference (Net) = -0.5, Standard Error of Mean 1.2

40. Other Pre Specified Outcome: Perceived Stress
Description: as for outcome 9
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale | -2.4 (1.3) | -0.1 (1.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.2, Mixed Models Analysis; Mean Difference (Net) = -2.3, Standard Error of Mean 1.8

41. Other Pre Specified Outcome: Exercise Self-Efficacy
Description: as for outcome 13
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -3.1 (4.9) | -6.8 (4.8)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.59, Mixed Models Analysis; Mean Difference (Net) = 3.7, Standard Error of Mean 6.9

42. Other Pre Specified Outcome: Weight-Related Quality of Life
Description: as for outcome 7
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale
  Total | 14.3 (2.5) | 13.4 (2.5)
  Physical Function | 12.4 (3.1) | 13.2 (3.1)
  Self Esteem | 20.0 (3.9) | 17.7 (3.9)
  Sexual Life | 13.3 (3.7) | 11.6 (3.6)
  Work | 12.1 (3.1) | 11.8 (3.1)
  Public Distress | 12.6 (2.7) | 7.6 (2.7)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Total; Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Net) = 0.9, Standard Error of Mean 3.5
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Physical Function; Test type: Superiority; p = 0.86, Mixed Models Analysis; Mean Difference (Net) = 0.8, Standard Error of Mean 4.4
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Self Esteem; Test type: Superiority; p = 0.87, Mixed Models Analysis; Mean Difference (Net) = 1.2, Standard Error of Mean 7.0
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Sexual Life; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Net) = 1.8, Standard Error of Mean 5.2
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Work; Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 4.4
Statistical Analysis 6: Comparison: BWL + BIAS vs Standard BWL; Public Distress; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = 5.0, Standard Error of Mean 3.8

43. Other Pre Specified Outcome: Eating Self-Efficacy
Description: as for outcome 15
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: scores on scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on scale | 8.3 (3.4) | 1.0 (3.4)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = 7.3, Standard Error of Mean 4.9

44. Other Pre Specified Outcome: Percent Weight Change
Description: Estimated mean change in percent weight change. Weight measured in kilograms (kg)
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: percent weight change
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
percent weight change | -3.1 (1.0) | -4.0 (1.0)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = 0.9, Standard Error of Mean 1.5

45. Other Pre Specified Outcome: Waist Circumference
Description: Estimated mean change in waist circumference (cm)
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: change in cm
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
change in cm | -4.4 (1.0) | -4.4 (1.0)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Net) = 0.0, Standard Error of Mean 1.5

46. Other Pre Specified Outcome: Blood Pressure
Description: as for outcome 19
Time Frame: Baseline to week 52
Measure: Mean (Standard Error); unit: change in mmHg
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
change in mmHg
  Systolic Blood Pressure | -5.7 (2.5) | -4.3 (2.5)
  Diastolic Blood Pressure | -1.1 (1.3) | -1.8 (1.3)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Systolic Blood Pressure; Test type: Superiority; p = 0.71, Mixed Models Analysis; Mean Difference (Net) = -1.4, Standard Error of Mean 3.6
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Diastolic Blood Pressure; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Net) = 0.7, Standard Error of Mean 1.9

47. Other Pre Specified Outcome: Body Esteem
Description: as for outcome 22
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.8 (0.1) | 0.4 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = 0.4, Standard Error of Mean 0.2

48. Other Pre Specified Outcome: Coping Behaviors in Response to Weight Stigma
Description: as for outcome 20
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Full Scale | -0.7 (0.1) | -0.6 (0.1)
  Negative Affect | -1.2 (0.1) | -0.8 (0.1)
  Maladaptive Eating | -0.6 (0.1) | -0.6 (0.1)
  Exercise Avoidance | -0.7 (0.3) | -0.6 (0.3)
  Healthy Lifestyle | -0.2 (0.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Full Scale; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Negative Affect; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Net) = -0.5, Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Maladaptive Eating; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.2
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Exercise Avoidance; Test type: Superiority; p = 0.74, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.4
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Healthy Lifestyle; Test type: Superiority; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.3

49. Other Pre Specified Outcome: Body Dissatisfaction
Description: as for outcome 24
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 0.5 (0.1) | 0.4 (0.1)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Net) = 0.2, Standard Error of Mean 0.2

50. Other Pre Specified Outcome: Anxiety
Description: as for outcome 30
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | -1.5 (0.9) | -0.3 (0.9)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Net) = -1.2, Standard Error of Mean 1.2

51. Other Pre Specified Outcome: Disordered Eating
Description: as for outcome 26
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Global | -0.4 (0.1) | -0.2 (0.1)
  Eating Restraint | 1.0 (0.3) | 0.7 (0.3)
  Eating Concern | -0.6 (0.2) | -0.3 (0.2)
  Weight Concern | -1.0 (0.2) | -0.7 (0.2)
  Shape Concern | -1.1 (0.2) | -0.7 (0.2)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Global; Test type: Superiority; p = 0.35, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Eating Restraint; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Eating Concern; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Net) = -0.3, Standard Error of Mean 0.3
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Weight Concern; Test type: Superiority; p = 0.18, Mixed Models Analysis; Mean Difference (Net) = -0.4, Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: BWL + BIAS vs Standard BWL; Shape Concern; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = -0.5, Standard Error of Mean 0.3

52. Other Pre Specified Outcome: Eating Behaviors
Description: as for outcome 28
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Dietary Restraint | 3.5 (0.9) | 3.2 (0.9)
  Disinhibition | -1.8 (0.5) | -1.2 (0.6)
  Hunger | -2.9 (0.6) | -0.7 (0.6)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Dietary Restraint; Test type: Superiority; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = 0.3, Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Disinhibition; Test type: Superiority; p = 0.45, Mixed Models Analysis; Mean Difference (Net) = -0.6, Standard Error of Mean 0.8
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Hunger; Test type: Superiority; p = 0.007, Mixed Models Analysis; Mean Difference (Net) = -2.2, Standard Error of Mean 0.8

53. Other Pre Specified Outcome: Self-Reported Self-Monitoring Behaviors
Description: as for outcome 34
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  Self-Reported Weighing | 0.9 (0.2) | 0.5 (0.2)
  Track Food/Drink | 0.8 (0.2) | 0.7 (0.2)
  Track Calories | 1.2 (0.3) | 1.3 (0.3)
  Track Activity | 0.8 (0.3) | 0.3 (0.3)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Self-Reported Weighing; Test type: Superiority; p = 0.23, Mixed Models Analysis; Mean Difference (Net) = 0.4, Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: BWL + BIAS vs Standard BWL; Track Food/Drink; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: BWL + BIAS vs Standard BWL; Track Calories; Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: BWL + BIAS vs Standard BWL; Track Activity; Test type: Superiority; p = 0.30, Mixed Models Analysis; Mean Difference (Net) = 0.4, Standard Error of Mean 0.5

54. Other Pre Specified Outcome: Treatment Acceptability Ratings
Description: To assess treatment acceptability, participants in both groups rated (1-7) the BWL treatment, as well as the stigma intervention (i.e., BIAS component) or recipe exchange, on how helpful they found each component of the program, how much they liked the components, and how much they learned new skills or information from each component. Scores for these three items were averaged (1-7) separately for the BWL treatment, BIAS component, and recipe exchange. Higher scores indicate greater treatment acceptability.
Time Frame: Week 26
Population: Participants randomized to the BWL + BIAS group did not receive (and thus did not rate) the recipe exchange component of treatment. Participants in the Standard BWL group did not receive (and did not rate) the BIAS treatment component.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale
  BWL component | 6.5 (0.9) | 6.3 (1.0)
  BIAS component: number analyzed (Participants) | 36 | 0
  BIAS component | 6.3 (1.0) |
  Recipe exchange: number analyzed (Participants) | 0 | 36
  Recipe exchange |  | 5.4 (1.5)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; BWL component; Test type: Superiority; p = 0.32, ANOVA

55. Other Pre Specified Outcome: Treatment Acceptability Ratings
Description: To assess treatment acceptability, participants rated (1-7) 5 items to indicate the extent to which they found the program (as a whole) to be helpful and acceptable, and how much they liked, were satisfied with, and would recommend the program to others. Scores are averaged 1-7, with higher scores indicating greater treatment acceptability.
Time Frame: Week 52
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BWL + BIAS | Standard BWL
Number analyzed (Participants) | 36 | 36
scores on a scale | 6.5 (0.6) | 6.2 (0.9)
Statistical Analysis 1: Comparison: BWL + BIAS vs Standard BWL; Test type: Superiority; p = 0.14, ANOVA

ADVERSE EVENTS:
Time Frame: Week 1 through week 26
Description: At each contact with participants, study personnel non-systematically collected information on any adverse events (AEs) self-reported by participants. In addition, AEs were systematically assessed at the scheduled assessments. AEs were documented by study staff in consultation with a nurse practitioner and/or physician. Serious adverse events (SAEs) were reported immediately to the study sponsor, Data and Safety Monitor, and the Institutional Review Board.
Arm/Group | BWL + BIAS | Standard BWL
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/36
Other Adverse Events (participants affected / at risk) | 3/36 | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BWL + BIAS (N=36) | Standard BWL (N=36)
Hypokalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BWL + BIAS (N=36) | Standard BWL (N=36)
Viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03572218/Prot_SAP_003.pdf